CLINICAL TRIAL: NCT04616651
Title: Patient-centered Development of the Cancer Support Community's Open to Options ®Chatbot Program Cancer Treatment Support in Partnership With the Cancer Support Community
Brief Title: Patient-centered Development of the Cancer Support Community's Open to Options ®Chatbot Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Cancer Support Community (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2020.083; HUM00179538 (Other: University of Michigan)
Record Dates: First submitted 2020-10-06; First posted 2020-11-05 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Cancer
Keywords: Chatbot; Open to Options (O2O)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Chatbot survey arm (Active Comparator): Participants will take the self-appraisal survey prior to interacting with the O2O program via the online Chatbot.
  Interventions: Behavioral: Online Survey; Behavioral: Chatbot prototype; Behavioral: Open to Options (O2O) Program
- Post-Chatbot survey arm (Experimental): Participants will take the self-appraisal survey after interacting with the O2O program via the online Chatbot. (This arm will also answer additional questions regarding participants' satisfaction with the O2O Chatbot.)
  Interventions: Behavioral: Online Survey; Behavioral: Chatbot prototype; Behavioral: Open to Options (O2O) Program

INTERVENTIONS:
Behavioral: Online Survey — Participants respond to online survey questions either before or after using the Chatbot O2O intervention.
  Other Names: Qualtrix Survey
Behavioral: Chatbot prototype — An online, automated, menu-based agent in which all responses are pre-programmed to be consistent with the existing O2O program. The chat-like responses help guide the participant through a process with the goal of developing a list of questions for their upcoming appointment with a cancer clinician. The session is meant to be completed in one sitting and estimated to take about 45 minutes to complete (including the pre- or post-intervention survey); however, if a participant stops in the middle, they may go back and complete the Chatbot session (or survey).
Behavioral: Open to Options (O2O) Program — Evidence-based program developed by Cancer Support Community that helps patients actively engage in their treatment decision process by preparing them for their upcoming appointments.

SUMMARY:
This study is designed to study the feasibility and acceptability of the Open to Options (O2O) Chatbot prototype. The O2O program is an existing patient support program with content currently delivered via in-person counseling with a trained mental health professional or via an existing web-based program (Let's Talk Treatment Options).The Chatbot is an automated, menu-based agent being developed in this study to extend the reach and accessibility of the O2O program via the Chatbot's "virtual coaching".

DETAILED DESCRIPTION:
This is a pilot study to assess feasibility and acceptability, and to gather preliminary data on how patients with a diagnosis of cancer appraise being prepared for their upcoming visit with a cancer specialist. Participants will be randomized to take a survey either before or after their Chatbot interaction. The surveys collect participants' self-appraisal regarding preparedness for their upcoming appointment with a cancer physician, cancer distress and cancer anxiety. The study will examine whether patients who take the survey after viewing the Chatbot feel more prepared for their upcoming appointment than those who take the survey before the Chatbot interaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cancer diagnosis
* Able to speak and read English, and willing to electronically consent
* Appointment with a Rogel Cancer Center cancer clinician within the next 3 weeks
* Patient must have a way to access the internet (includes mobile phone)

Exclusion Criteria:

* Age <18 years
* Inability to speak or read English
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of Integrating Chatbot in Clinic | At the time of scheduling an appointment with cancer physician; one day
  The feasibility of integrating an Open to Options (O2O) Chatbot into the clinical workflow, assessed by the number of patients who accept the invitation to receive more information about the study, among all those invited.
Acceptability - Reach | Baseline (Before appointment with cancer physician); up to approximately 3 weeks after scheduling appointment
  Assessed by the number of patients who log-in to the O2O Chatbot program and create an account, among all those who accepted the invitation to receive information.
Acceptability - Uptake | Baseline (Before appointment with cancer physician); up to approximately 3 weeks after scheduling appointment
  Assessed by the number of patients who proceed to view the full Chatbot prototype and generate a summary, among all those who created an account.
Acceptability - Mean Satisfaction Scores | Baseline (Before appointment with cancer physician); up to approximately 3 weeks after scheduling appointment
  Post-Intervention Survey Group only: In addition to the survey given to all participants, the post-intervention survey group will answer 6 questions about their perception of the Chatbot prototype. Each of the 6 questions will be scored on a scale from 1 (strongly disagree) to 5 (strongly agree). Investigators will calculate the mean value (and Standard Deviation) on a 1-5 scale for each question.
Acceptability - Percent of Participants with High Satisfaction Scores | Baseline (Before appointment with cancer physician); up to approximately 3 weeks after scheduling appointment
  Post-Intervention Survey Group only: In addition to the survey given to all participants, the post-intervention survey group will answer 6 questions about their perception of the Chatbot prototype. Each of the 6 questions will be scored on a scale from 1 (strongly disagree) to 5 (strongly agree). For each of the six questions, investigators will calculate the percentage of participants who strongly agree.

OTHER OUTCOMES:
Mean Patient-reported Appraisal Outcomes | Baseline (Before appointment with cancer physician); up to approximately 3 weeks after scheduling appointment
  Mean values of the following 5 self-appraisals:
  * Cancer related distress [scale from 0 (none) to 10 (extreme)]
  * Cancer diagnosis anxiety [scale from 0 (none) to 10 (extreme)]
  * Self-efficacy for question asking [scale from 0 (not at all confident) to 10 (extremely confident)]
  * Decision preparedness [scale from 1 (not at all) to 5 (a great deal)]
  * Decision self-efficacy [scale from 0 (not at all confident) to 4 (very confident)]
  The mean values will be compared by group (pre- vs. post-intervention survey group) using t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hawley, PhD, MPH, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No